CLINICAL TRIAL: NCT07360314
Title: A Phase 1, 2-Part, Multicenter, Open-Label, First-in-Human Study of the Anti-Ly6E Exatecan Antibody-Drug Conjugate M7437 in Participants With Advanced Solid Tumors
Brief Title: Anti-Ly6E Exatecan ADC M7437 in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MS743701_0001; 176325 (Other: IND); 2025-523232-39-00 (EU CTIS Number); NCT07311603 (obsolete NCT alias)
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: Ly6E expression; Topoisomerase I inhibitor (TOP1i); NSCLC; Breast cancer; Gastric cancer; Head and neck squamous cell carcinoma; Ovarian cancer; Pancreatic ductal adenocarcinoma; Systemic antibody-drug conjugate therapy (ADC) therapy
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose-escalation Cohort (Experimental)
  Interventions: Drug: M7437
- Part 2: Dose-Expansion Cohort (Experimental)
  Interventions: Drug: M7437

INTERVENTIONS:
Drug: M7437 — Participants will receive M7437 as an intravenous infusion at a dose corresponding to their assigned cohort. Dose escalation will occur between cohorts, with 3-4 participants enrolled at each dose level before proceeding to the next higher dose.
  Arms: Part 1: Dose-escalation Cohort
Drug: M7437 — Participants will receive M7437 at a dose that was determined as recommended dose for expansion (RDE) in Part 1.
  Arms: Part 2: Dose-Expansion Cohort

SUMMARY:
The purpose of this first-in-human (FIH) study is to evaluate the safety, tolerability, Pharmacokinetics (PK), and preliminary clinical activity of M7437 in participants with locally advanced or metastatic solid tumors with known Ly6E expression, including non-small cell lung cancer (NSCLC), triple-negative breast cancer (TNBC), epithelial ovarian carcinoma (EOC), squamous cell carcinoma of the head and neck (SCCHN), pancreatic ductal adenocarcinoma (PDAC), and gastric cancer (GC).

ELIGIBILITY:
Inclusion Criteria:

* Participants have histologically proven advanced solid tumors with known prevalent and high Ly6E expression, Disease characteristic: Participants should have an unresectable locally advanced or metastatic solid tumor that is refractory to standard therapies, or have no standard therapies, or for which no standard therapy is judged appropriate by the Investigator.

For each tumor type, participants have received prior lines of therapy, where locally available:

* Non-small cell lung cancer (nonsquamous or squamous)
* Triple-negative breast cancer
* Squamous cell carcinoma of head and neck
* Pancreatic ductal adenocarcinoma
* Gastric cancer
* Epithelial ovarian cancer

  * Participants with ECOG Performance Status (ECOG) less than and equal to (<=) 1
  * Participants must have blood, liver, and kidney function within safe levels.
  * Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* Participant has a history of another malignancy within 3 years before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, benign prostate neoplasm/hyperplasia, or malignancy that in the opinion of the Investigator, with concurrence with the Sponsor's Medical Monitor, is considered cured with minimal risk of recurrence within 3 years before the date of enrollment). History of hematopoietic allogenic transplantation.
* Participants with known brain metastases, except those meeting both of the following criteria:

  1. All brain metastases have been treated locally and are clinically stable for at least 4 weeks prior to the start of treatment.
  2. No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable).
* Participants with diarrhea (liquid stool) or ileus Grade more than (>) 1 within 1 week of Cycle1Day1.
* Participants with active chronic inflammatory bowel disease and/or bowel obstruction.
* Participants with history of serious gastrointestinal bleeding within 3 months of Cycle1Day1.
* Other protocol defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-09-20 (Estimated); Study Completion 2029-03-28 (Estimated)

PRIMARY OUTCOMES:
Dose-escalation Cohort: Occurences of Dose Limiting Toxicities (DLTs) | DLT period is 21 days (cycle 1)
Dose-escalation Cohort: Number of Participants With Treatment-Emergent Adverse Event (TEAEs) and Adverse Event (AEs) | Up to end of Part 1 of study (approximately 1 year 8 months)

SECONDARY OUTCOMES:
Dose-escalation Cohort: Plasma Concentration of M7437 | Cycle 1 Day 1: Pre-dose, 0.25, 6, 24, 96, 168 and 336 hours post-dose; Cycle 3 Day 1: Pre-dose, 0.25, 6 and 168 hours post-dose; Pre-dose at Day 1 of Cycles 2, 4, 6, 8 until end of treatment (approximately 1 year 8 months) (Each Cycle length=21 days)
Dose-escalation Cohort: Overall Response (OR) According to Response Evaluation Criteria inSolid Tumor (RECIST) version 1.1 criteria as Assessed by Investigator | From the date of first documented complete response (CR) or partial response (PR), whichever occurs first, until the first documented disease recurrence or progressive disease (PD) (assessed upto [approximately 1 year 8 months])
Change From The Baseline Qtc (Δqtc) At Predefined Timepoints Based on Triplicate Electrocardiogram (ECG) Measurements | Baseline, Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 5, Cycle 1 Day 8, Cycle 2 Day 1, Cycle 3 Day 1 (each cycle is of 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (8):
- United States (4):
  - Yale University - Yale University School of Medicine, New Haven, Connecticut
  - Carolina BioOncology Institute, LLC - Cancer Therapy and Research Center, Huntersville, North Carolina
  - NEXT Houston, Galveston, Texas
  - NEXT Oncology - PARENT, San Antonio, Texas
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto
  - BC Cancer - Vancouver - BC Cancer Agency, Vancouver
- National Cancer Center Hospital, Tokyo, Japan
- NEXT Madrid - Hospital Universitario Quironsalud Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS743701_0001
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html